CLINICAL TRIAL: NCT02904486
Title: Effectiveness of Modified Health Belief Model Based Intervention to Reduce Body Mass
Brief Title: Effectiveness of Modified Health Belief Model Based Intervention to Reduce Body Mass Index
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Waraporn Khumros, Department of Preventive and Social Medicine Faculty of Medicine, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AUI-9959
Record Dates: First submitted 2016-09-09; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- change behavior (Experimental): Modified Health Belief Model Based Intervention and study health topic in classroom to change behavior for Reduce Body Mass Index for Age in Overweight Junior High School Students.
  Interventions: Behavioral: change behavior
- lifestyle behavior (Experimental): study health topic in classroom to change behavior for Reduce Body Mass Index for Age in Overweight Junior High School Students.
  Interventions: Behavioral: change behavior

INTERVENTIONS:
Behavioral: change behavior — Modified Health Belief Model Based Intervention to Reduce Body Mass Index for Age
  Other Names: change behavior intervention

SUMMARY:
The purpose of this study is to Effectiveness of Modified Health Belief Model Based Intervention to Reduce Body Mass Index for Age in Overweight Junior High School Students.

DETAILED DESCRIPTION:
The purpose of this study is to Effectiveness of Modified Health Belief Model Based Intervention to change behavior to Reduce Body Mass Index for Age in Overweight Junior High School Students.

ELIGIBILITY:
Inclusion Criteria:

* junior High School Students
* age 12 - 15 years
* bmi for age ≥ median +1 SD
* Read and write Thai Language
* Agree to participate voluntarily .

Exclusion Criteria:

* students with medical conditions diagnosed by a physician and a barrier to participation .

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 232 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index | 6 month
  Modified Health Belief Model Based Intervention to Reduce Body Mass Index for Age in Overweight Junior High School Students durationof program 6 month

SECONDARY OUTCOMES:
Heath literacy for obesity in Junior High School Students. | 6 month
  assessment to Heath literacy for obesity in Junior High School Students by questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: waraporn khumros, Ph.D study, Principal Investigator — Chulalongkorn University

IPD SHARING:
Plan to Share IPD: Yes